CLINICAL TRIAL: NCT01225393
Title: A Phase II, Randomized, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of MLTA3698A in Combination With a Disease-Modifying Anti-Rheumatic Drug (DMARD) Compared With Adalimumab in Combination With a DMARD in Patient With Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of MLTA3698A in Combination With a Disease-Modifying Anti-Rheumatic Drug (DMARD) Compared With Adalimumab in Combination With a DMARD in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT4864g; GA00932 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — pateclizumab; Adalimumab; Leflunomide; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental)
  Interventions: Drug: MLTA3698A; Drug: leflunomide; Drug: methotrexate
- B (Active Comparator)
  Interventions: Drug: adalimumab; Drug: leflunomide; Drug: methotrexate; Drug: placebo
- C (Placebo Comparator)
  Interventions: Drug: leflunomide; Drug: methotrexate; Drug: placebo

INTERVENTIONS:
Drug: MLTA3698A — Subcutaneous repeating dose
  Arms: A
Drug: adalimumab — Subcutaneous repeating dose
  Arms: B
Drug: leflunomide — Stable dose if not on methotrexate
Drug: methotrexate — Stable dose if not on leflunomide
Drug: placebo — Subcutaneous repeating dose
  Arms: B; C

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled, parallel-group, multicenter study enrolling patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the 1987 revised ACR Criteria for the Classification of RA for at least 6 months prior to screening
* Positive for rheumatoid factor or anti-cyclic citrullinated peptide (CCP) antibody, or both
* Active disease, defined as: CRP >= 1.0 mg/dL; swollen joint count >= 6 (66 joint count); tender joint count >= 6 (68 joint count)
* Previous inadequate clinical response to at least one disease-modifying anti-rheumatic drug (DMARD) consisting of either methotrexate (MTX) or leflunomide (LFU)
* For patients currently receiving corticosteroids: Treatment at a stable dose during last 4 weeks prior to screening
* For patients currently receiving non-steroidal anti-inflammatory drugs (NSAIDs): Treatment at a stable dose during last 4 weeks prior to screening
* For patients currently receiving sulfasalazine or anti-malarials: Treatment initiated and continued for at least the last 6 months prior to screening and on a stable dose
* For patients of reproductive potential (males and females): Willing to use a highly effective birth control method for the duration of the study according to local guidelines

Exclusion Criteria:

* Pregnant, planning to become pregnant during the study, or breastfeeding
* Clinically significant abnormal laboratory values or abnormal ECG or vital signs
* History of anaphylactic reactions
* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis, or Felty's syndrome), however patients with secondary Sjogren's syndrome are eligible for the study
* History of or current inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthritis, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, or other overlap syndrome)
* Current or recent (within 4 weeks prior to screening) infection, including signs, symptoms or serology of any infection, including HIV, hepatitis B or C, tuberculosis
* Administration of a live, attenuated vaccine within 1 month before dosing or anticipation that such a live attenuated vaccine will be required during the study
* Previous treatment with anti-TNF biologics or other biologic agents, including anti-CD20-directed therapy (e.g. rituximab), anti-IL6-directed therapy (e.g. tocilizumab), or T cell-directed therapy (e.g. abatacept)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Baseline change in disease activity, assessed as the Disease Activity Score (DAS28) and erythrocyte sedimentation rate, or DAS28-(4)-ESR | Day 85
Incidence and severity of adverse events and clinical laboratory abnormalities as a measure of safety and tolerability of MLTA3698A | Length of study (through Day 85)

SECONDARY OUTCOMES:
ACR20 response rate (the proportion of patients in each treatment group meeting the American College of Rheumatology 20% responder criteria [ACR20] for their average response ) | Day 85
ACR50 response rate (the proportion of patients in each treatment group meeting the American College of Rheumatology 50% responder criteria [ACR50] for their average response ) | Day 85
ACR70 response rate (the proportion of patients in each treatment group meeting the American College of Rheumatology 70% responder criteria [ACR70] for their average response) | Day 85
Tender joint count | Day 85
Swollen joint count | Day 85
Investigator Global Assessment of Disease Activity | Day 85
Patient Global Assessment of Pain and Disease Activity | Day 85
Health Assessment Questionnaire Disability Index | Day 85
Patient's Global Health or Short Form Health Survey (SF-36) | Day 85
European League Against Rheumatism response rate | Day 85
Serum C-reactive protein levels | Day 85
Erythrocyte sedimentation rate | Day 85

CONTACTS AND LOCATIONS:
Overall Officials: John C. Davis, Jr., M.D., M.P.H., Study Director — Genentech, Inc.
Locations (52):
- United States (14):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Peoria, Arizona
  - Los Angeles, California
  - Upland, California
  - Ormond Beach, Florida
  - Lexington, Kentucky
  - Kalamazoo, Michigan
  - Flowood, Mississippi
  - Reno, Nevada
  - Charleston, South Carolina
  - San Antonio, Texas
  - Chesapeake, Virginia
  - Clarksburg, West Virginia
- Sofia, Bulgaria
- Santiago, Chile
- Germany (8):
  - Bad Nauheim
  - Berlin
  - Cologne
  - Erfurt
  - Freiburg im Breisgau
  - Herne
  - Kiel
  - Zerbst
- Hungary (4):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Veszprém
- Mexico (8):
  - Culiacán
  - Guadalajara
  - León
  - Mexicali
  - Mexico City
  - Mérida
  - México
  - Monterrey, NL
- Peru (2):
  - Lima
  - San Isidro
- Poland (6):
  - Bialystok
  - Elblag
  - Kościan
  - Krakow
  - Lublin
  - Warsaw
- Romania (4):
  - Baia Mare
  - Bucharest
  - Cluj-Napoca
  - Galati
- Spain (4):
  - Torrelavega, Cantabria
  - A Coruña, La Coruña
  - Seville, Sevilla
  - S. Cristobal de La Laguna, Tenerife

REFERENCES:
- [Derived] Kennedy WP, Simon JA, Offutt C, Horn P, Herman A, Townsend MJ, Tang MT, Grogan JL, Hsieh F, Davis JC. Efficacy and safety of pateclizumab (anti-lymphotoxin-alpha) compared to adalimumab in rheumatoid arthritis: a head-to-head phase 2 randomized controlled study (The ALTARA Study). Arthritis Res Ther. 2014 Oct 30;16(5):467. doi: 10.1186/s13075-014-0467-3. PMID 25359150